CLINICAL TRIAL: NCT03955588
Title: Demonstration Trial on Replacement of Cytogenetics by Array Comparative Genomic Hybridisation (aCGH) in Prenatal Diagnosis
Brief Title: Replacement of Cytogenetics by aCGH in Prenatal Diagnosis
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Hui Pui-Wah, Prinicipal Investigator, The University of Hong Kong
Other Study IDs: UW 14-465
Record Dates: First submitted 2019-05-07; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Prenatal Diagnosis
Keywords: Cytogenetics; aCGH; Prenatal Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing invasive prenatal diagnostic procedures: For women requiring invasive prenatal diagnosis by chorionic villus sampling or amniocentesis, they will be offered the options of having either conventional cytogenetics or aCGH.
  Interventions: Diagnostic Test: aCGH

INTERVENTIONS:
Diagnostic Test: aCGH
  Other Names: conventional cytogenetics

SUMMARY:
Conventional cytogenetics has been the gold standard for chromosomal analysis in prenatal diagnosis. It allows a microscopic examination for any structural abnormalities of chromosome with a turn-around time of 2 to 3 weeks and it is also labour intensive. Array comparative genome hybridisation (aCGH) provides a platform for a higher resolution analysis of chromosomal aberrations in a shorter period of time. The effectiveness of its application in prenatal diagnosis has been examined. The main clinical limitation lies on the difficult interpretation of certain copy number variants (CNV). Our previous study has demonstrated an increase diagnostic yield of 3.2% using aCGH over conventional cytogenetics in the first-tier test study and by 6% as a further test in a cohort of fetuses with ultrasound abnormality and normal karyotype findings. This finding were consistent with the overall reported of 5.2% to 10% increased detection rate by other studies. Various authorities have also approved the use of aCGH as an adjunct diagnostic tool in prenatal cases with fetal ultrasound abnormalities.

The presence study aims to demonstrate the clinical acceptability on the use of aCGH to replace cytogenetics in prenatal diagnosis. For patients requiring invasive prenatal diagnosis by chorionic villus sampling or amniocentesis, they will be offered the options of having either conventional cytogenetics or aCGH. A standard unbiased counselling procedure will be performed by well trained midwives. For patients opting for conventional cytogenetics, the current procedure of karyotyping will be performed. For those opting for aCGH, a quantitative fluorescent Polymerase Chain Reaction (PCR) will be performed first to exclude common aneuploidies and triploidies. aCGH will be arranged for those with normal PCR results and conventional cytogenetics will be reserved for visualization of clinically significant CNVs.

All patients will be asked to complete the same questionnaire that has been adopted for the study on "Questionnaire survey on Knowledge and Acceptance on Application of whole genome array Comparative Genomic Hybridisation (aCGH) in Prenatal Diagnosis".

DETAILED DESCRIPTION:
Conventional cytogenetics has been the gold standard for chromosomal analysis in prenatal diagnosis. It allows a microscopic examination for any structural abnormalities of chromosome with a turn-around time of 2 to 3 weeks and it is also labour intensive. Array comparative genome hybridisation (aCGH) provides a platform for a higher resolution analysis of chromosomal aberrations in a shorter period of time. The effectiveness of its application in prenatal diagnosis has been examined (Callaway, Shaffer, Chitty, Rosenfeld, & Crolla, 2013). The main clinical limitation lies on the difficult interpretation of certain copy number variants (CNV). Our previous study has demonstrated an increase diagnostic yield of 3.2% using aCGH over conventional cytogenetics in the first-tier test study and by 6% as a further test in a cohort of fetuses with ultrasound abnormality and normal karyotype findings (Kan et al., 2014). This finding were consistent with the overall reported of 5.2% to 10% increased detection rate by other studies (de Wit et al., 2014; Hillman et al., 2013; Hillman et al., 2011). Various authorities have also approved the use of aCGH as an adjunct diagnostic tool in prenatal cases with fetal ultrasound abnormalities (American College of Obstetricians & Gynecologists, 2013; Novelli et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

All pregnant women requiring chorionic villus sampling or amniocentesis at Tsan Yuk Hospital

Exclusion Criteria:

Patients who cannot read or understand Chinese or English

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women who require invasive prenatal diagnosis will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
The preference of aCGH to conventional cytogenetics | At the time of recruitment
  Proportion of subjects choosing aCGH

SECONDARY OUTCOMES:
Cost-effectiveness analysis of chromosomal microarray as primary test for prenatal diagnosis in Hong Kong | After completion of the aCGH for the last recruited subject in 2016
  Laboratory workflow and cost of replacing conventional karyotype by aCGH are compared. The cost-effectiveness analysis is based on the diagnostic rate (number of diagnoses made/ sample size) as a measure of outcome effectiveness.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists Committee on Genetics. Committee Opinion No. 581: the use of chromosomal microarray analysis in prenatal diagnosis. Obstet Gynecol. 2013 Dec;122(6):1374-7. doi: 10.1097/01.AOG.0000438962.16108.d1. PMID 24264715
- [Background] Callaway JL, Shaffer LG, Chitty LS, Rosenfeld JA, Crolla JA. The clinical utility of microarray technologies applied to prenatal cytogenetics in the presence of a normal conventional karyotype: a review of the literature. Prenat Diagn. 2013 Dec;33(12):1119-23. doi: 10.1002/pd.4209. Epub 2013 Sep 8. PMID 23983223
- [Background] de Wit MC, Srebniak MI, Govaerts LC, Van Opstal D, Galjaard RJ, Go AT. Additional value of prenatal genomic array testing in fetuses with isolated structural ultrasound abnormalities and a normal karyotype: a systematic review of the literature. Ultrasound Obstet Gynecol. 2014 Feb;43(2):139-46. doi: 10.1002/uog.12575. PMID 23897843
- [Background] Hillman SC, McMullan DJ, Hall G, Togneri FS, James N, Maher EJ, Meller CH, Williams D, Wapner RJ, Maher ER, Kilby MD. Use of prenatal chromosomal microarray: prospective cohort study and systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2013 Jun;41(6):610-20. doi: 10.1002/uog.12464. Epub 2013 May 7. PMID 23512800
- [Background] Hillman SC, Pretlove S, Coomarasamy A, McMullan DJ, Davison EV, Maher ER, Kilby MD. Additional information from array comparative genomic hybridization technology over conventional karyotyping in prenatal diagnosis: a systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2011 Jan;37(1):6-14. doi: 10.1002/uog.7754. PMID 20658510
- [Background] Kan AS, Lau ET, Tang WF, Chan SS, Ding SC, Chan KY, Lee CP, Hui PW, Chung BH, Leung KY, Ma T, Leung WC, Tang MH. Whole-genome array CGH evaluation for replacing prenatal karyotyping in Hong Kong. PLoS One. 2014 Feb 5;9(2):e87988. doi: 10.1371/journal.pone.0087988. eCollection 2014. PMID 24505343
- [Background] Novelli A, Grati FR, Ballarati L, Bernardini L, Bizzoco D, Camurri L, Casalone R, Cardarelli L, Cavalli P, Ciccone R, Clementi M, Dalpra L, Gentile M, Gelli G, Grammatico P, Malacarne M, Nardone AM, Pecile V, Simoni G, Zuffardi O, Giardino D. Microarray application in prenatal diagnosis: a position statement from the cytogenetics working group of the Italian Society of Human Genetics (SIGU), November 2011. Ultrasound Obstet Gynecol. 2012 Apr;39(4):384-8. doi: 10.1002/uog.11092. PMID 22262341